CLINICAL TRIAL: NCT04068181
Title: Phase 2 Study of Talimogene Laherparepvec in Combination With Pembrolizumab in Subjects With Unresectable/Metastatic Stage IIIB-IVM1d Melanoma Who Have Progressed on Prior Anti PD-1 Based Therapy
Brief Title: Talimogene Laherparepvec With Pembrolizumab in Melanoma Following Progression on Prior Anti-PD-1 Based Therapy (MASTERKEY-115) (Mk-3475-A07/KEYNOTE-A07).
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20180115; 2019-001906-61 (EudraCT Number)
Record Dates: First submitted 2019-08-22; First posted 2019-08-28 (Actual); Results first posted 2022-09-09 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-11

CONDITIONS: Melanoma
Keywords: Melanoma; Talimogene Laherparepvec; Pembrolizumab; Oncolytic immunotherapy; Anti-PD-1; Checkpoint inhibitor; MASTERKEY-115
MeSH Terms: conditions — Melanoma | interventions — talimogene laherparepvec; pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 - Locally Recurrent/Metastatic - Primary Resistance (Experimental): Includes participants who received anti-PD1 therapy in the locally recurrent/metastatic setting and experienced a best overall response of disease progression or stable disease prior to confirmed disease progression.
  Participants will receive talimogene laherparepvec at an initial dose of up to 4.0 mL of 10^6 plaque-forming units (PFU)/mL on Day 1. Subsequent doses of up to 4.0 mL of 10^8 PFU/mL will be administered every 3 weeks for up to 35 cycles in total. Participants will also receive pembrolizumab at a dose of 200 mg every 3 weeks for up to 35 cycles.
  Interventions: Drug: Talimogene laherparepvec; Drug: Pembrolizumab
- Cohort 2 - Locally Recurrent/Metastatic - Acquired Resistance (Experimental): Includes participants who received anti-PD-1 therapy in the locally recurrent/metastatic setting and experienced confirmed disease progression following a complete or partial response on anti-PD-1 therapy.
  Participants will receive talimogene laherparepvec at an initial dose of up to 4.0 mL of 10^6 plaque-forming units (PFU)/mL on Day 1. Subsequent doses of up to 4.0 mL of 10^8 PFU/mL will be administered every 3 weeks for up to 35 cycles in total. Participants will also receive pembrolizumab at a dose of 200 mg every 3 weeks for up to 35 cycles.
  Interventions: Drug: Talimogene laherparepvec; Drug: Pembrolizumab
- Cohort 3 - Adjuvant Setting -Disease Free Interval < 6 months (Experimental): Includes participants who received anti-PD-1 therapy in the adjuvant setting and experienced confirmed disease progression following a disease-free interval of < 6 months after starting the adjuvant anti-PD-1 therapy.
  Participants will receive talimogene laherparepvec at an initial dose of up to 4.0 mL of 10^6 plaque-forming units (PFU)/mL on Day 1. Subsequent doses of up to 4.0 mL of 10^8 PFU/mL will be administered every 3 weeks for up to 35 cycles in total. Participants will also receive pembrolizumab at a dose of 200 mg every 3 weeks for up to 35 cycles.
  Interventions: Drug: Talimogene laherparepvec; Drug: Pembrolizumab
- Cohort 4 - Adjuvant Setting -Disease Free Interval ≥ 6 months (Experimental): Includes participants who received anti PD-1 therapy in the adjuvant setting and experienced confirmed disease progression following a disease-free interval of ≥ 6 months after starting the adjuvant PD-1 inhibitor.
  Participants will receive talimogene laherparepvec at an initial dose of up to 4.0 mL of 10^6 plaque-forming units (PFU)/mL on Day 1. Subsequent doses of up to 4.0 mL of 10^8 PFU/mL will be administered every 3 weeks for up to 35 cycles in total. Participants will also receive pembrolizumab at a dose of 200 mg every 3 weeks for up to 35 cycles.
  Interventions: Drug: Talimogene laherparepvec; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Talimogene laherparepvec — Intralesional injection into injectable cutaneous, subcutaneous and nodal legions.
Drug: Pembrolizumab — Intravenous (IV) infusion.

SUMMARY:
This is a phase 2, open-label, single-arm, multicenter clinical trial designed to evaluate the efficacy and safety of talimogene laherparepvec in combination with pembrolizumab following disease progression on prior anti-programmed cell death protein (anti-PD-1) therapy in unresectable/metastatic melanoma (stage IIIB-IVM1d) or prior anti-PD-1 therapy in the adjuvant setting. Subjects will be treated with talimogene laherparepvec and pembrolizumab until confirmed complete response, disappearance of all injectable lesions, documented confirmed disease progression per modified immune-related Response Criteria simulating Response Evaluation Criteria in Solid Tumors (irRC-RECIST), intolerance of study treatment, or 102 weeks from the first dose of talimogene laherparepvec and/or pembrolizumab, whichever occurs first.

ELIGIBILITY:
Key Inclusion Criteria:

* Age ≥ 18 years with histologically confirmed diagnosis of stage IIIB to IVM1d melanoma and for whom surgery is not recommended. Subjects with stage IVM1d disease may be enrolled with up to 3 cerebral metastases, provided that all lesions have been adequately treated with stereotactic radiation therapy, craniotomy, or gamma knife therapy, with no evidence of progression and not requiring steroids for at least 2 months prior to enrollment.
* Subjects must have measurable disease and be a candidate for intralesional therapy administration into cutaneous, subcutaneous, or nodal lesions.
* Subjects must have had prior treatment (for at least 2 to 3 consecutive cycles within an 8 week period) with a PD-1 inhibitor and have confirmed disease progression (as defined by RECIST v1.1 criteria). The anti-PD-1 therapy must be the immediate prior line of therapy before enrollment and subjects with disease progression on more than 1 line of anti-PD-1 therapy are not eligible.
* ECOG performance status of 0 or 1.
* Adequate hematologic, renal, hepatic, and coagulation function.

Key Exclusion Criteria:

* Subjects considered by the investigator to have rapid clinical progression due to melanoma
* Subjects with prior treatment and disease progression on more than 1 line of anti-PD-1 therapy
* Stage IVM1d subjects must not have greater than 3 cerebral melanoma metastases, or clinically active cerebral melanoma metastases requiring therapy, and/or carcinomatous meningitis regardless of clinical stability.
* Primary uveal or mucosal melanoma, history or evidence of melanoma associated with immunodeficiency states or history of other malignancy within the past 3 years.
* Subjects must not have history or evidence of symptomatic autoimmune glomerulonephritis, vasculitis, or other symptomatic autoimmune disease, or active autoimmune disease or syndrome requiring systemic treatment in the past 2 years (ie, with use of disease modifying agents, steroids or immunosuppressive agents) except vitiligo or resolved childhood asthma/atopy, or evidence of clinically significant immunosuppression.
* Subjects may not have been previously treated with talimogene laherparepvec or any other oncolytic virus.
* Subjects must not have active herpetic skin lesions or prior complications of herpetic infection and must not require intermittent or chronic treatment with an antiherpetic drug (eg, acyclovir), other than intermittent topical use.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2021-08-19 (Actual); Study Completion 2024-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (46):
- United States (10):
  - Sansum Clinic, Santa Barbara, California
  - Medical Oncology Hematology Consultants Helen F Graham Cancer Center, Newark, Delaware
  - University of Florida Health Cancer Center at Orlando Health, Orlando, Florida
  - University of Louisville James Graham Brown Cancer Center, Louisville, Kentucky
  - Allina Health Systems dba Virginia Piper Cancer Institute, Fridley, Minnesota
  - New York Oncology Hematology, PC, Albany, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Texas Oncology Austin Central, Austin, Texas
  - Baylor Scott and White Research Institute, Dallas, Texas
  - United States Oncology Regulatory Affairs Corporate Office, The Woodlands, Texas
- Australia (5):
  - Melanoma Institute Australia, North Sydney, New South Wales
  - Tasman Oncology Research, Southport, Queensland
  - The Queen Elizabeth Hospital, Woodville South, South Australia
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - The Alfred Hospital, Melbourne, Victoria
- Canada (3):
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
  - CHU de Quebec-Universite Laval, Québec, Quebec
- France (6):
  - Centre Hospitalier Universitaire de Bordeaux - HÃ´pital Saint AndrÃ©, Bordeaux
  - Centre Hospitalier Universitaire de Grenoble - Hopital Nord Michallon, Grenoble
  - Centre Hospitalier Universitaire de Nantes, HÃ´pital HÃ´tel Dieu, Nantes
  - Hopital Saint Louis, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Gustave Roussy, Villejuif
- Germany (4):
  - UniversitÃ¤tsklinikum Carl Gustav Carus der Technischen UniversitÃ¤t Dresden, Dresden
  - Medizinische Hochschule Hannover, Hanover
  - UniversitÃ¤tsklinikum Regensburg, Regensburg
  - UniversitÃ¤tsklinikum TÃ¼bingen, TÃ¼bingen
- Greece (3):
  - General Hospital of Athens Laiko, Athens
  - University Hospital of Ioannina, Ioannina
  - Bioclinic of Thessaloniki, Thessaloniki
- Italy (3):
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII, Bergamo
  - IRCCS - Istituto Romagnolo per lo Studio dei Tumori (IRST) "Dino Amadori", Meldola FC
  - IRCCS Istituto Europeo di Oncologia, Milan
- Netherlands (2):
  - Nederlands Kanker Instituut, Antoni van Leeuwenhoekziekenhuis, Amsterdam
  - Erasmus Medisch Centrum, Rotterdam
- Poland (3):
  - Uniwersyteckie Centrum Kliniczne Centrum Medycyny Nieinwazyjnej, Gdansk
  - Szpital Kliniczny im Heliodora Swiecickiego Uniwersytetu Medycznego im Karola Marcinkowskiego w Pozn, Poznan
  - Narodowy Instytut Onkologii im Marii Sklodowskiej-Curie â€" Panstwowy Instytut Badawczy, Warsaw
- Spain (5):
  - Hospital Clinico Universitario Virgen de la Victoria, Málaga, AndalucÃ-a
  - Onkologikoa, Donostia / San Sebastian, PaÃ-s Vasco
  - Hospital Universitari Vall d Hebron, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Madrid Sanchinarro, Madrid
- United Kingdom (2):
  - Guys Hospital, London
  - Royal Marsden Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- [Background] Robert C, Gastman B, Gogas H, Rutkowski P, Long GV, Chaney MF, Joshi H, Lin YL, Snyder W, Chesney JA. Open-label, phase II study of talimogene laherparepvec plus pembrolizumab for the treatment of advanced melanoma that progressed on prior anti-PD-1 therapy: MASTERKEY-115. Eur J Cancer. 2024 Aug;207:114120. doi: 10.1016/j.ejca.2024.114120. Epub 2024 May 15. PMID 38870745
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 72 participants were enrolled at 28 centers in Australia, Canada, France, Germany, Greece, Italy, the Netherlands, Poland, Spain and the United States from 22 January 2020 to 26 February 2024.
Pre-assignment Details: Participants must have received prior anti-programmed cell death protein (anti-PD-1) therapy for at least 2 to 3 consecutive cycles within an 8-week period and have disease progression as defined by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria. The anti-PD-1 therapy must have been the immediate prior line of therapy before enrollment, and participants with disease progression on more than 1 line of anti-PD-1 therapy were not eligible.
Groups:
- Cohort 1 - Locally Recurrent/Metastatic - Primary Resistance: Included participants who received anti-PD-1 therapy in the locally recurrent/metastatic setting and experienced a best overall response of disease progression or stable disease prior to confirmed disease progression.
  Participants received talimogene laherparepvec at an initial dose of up to 4.0 mL of 10^6 plaque-forming units (PFU)/mL by intralesional injection into injectable cutaneous, subcutaneous and nodal legions on Day 1. Subsequent doses of up to 4.0 mL of 10^8 PFU/mL were administered every 3 weeks for up to 35 cycles in total. Participants also received pembrolizumab at a dose of 200 mg as an intravenous (IV) infusion every 3 weeks for up to 35 cycles.
- Cohort 2 - Locally Recurrent/Metastatic - Acquired Resistance: Included participants who received anti-PD-1 therapy in the locally recurrent/metastatic setting and experienced confirmed disease progression following a complete or partial response on anti-PD-1 therapy.
  Participants received talimogene laherparepvec at an initial dose of up to 4.0 mL of 10^6 PFU/mL by intralesional injection into injectable cutaneous, subcutaneous and nodal legions on Day 1. Subsequent doses of up to 4.0 mL of 10^8 PFU/mL were administered every 3 weeks for up to 35 cycles in total. Participants also received pembrolizumab at a dose of 200 mg as an IV infusion every 3 weeks for up to 35 cycles.
- Cohort 3 - Adjuvant Setting - Disease Free Interval < 6 Months: Included participants who received anti-PD-1 therapy in the adjuvant setting and experienced confirmed disease progression following a disease-free interval of < 6 months after starting the adjuvant anti-PD-1 therapy.
  Participants received talimogene laherparepvec at an initial dose of up to 4.0 mL of 10^6 PFU/mL by intralesional injection into injectable cutaneous, subcutaneous and nodal legions on Day 1. Subsequent doses of up to 4.0 mL of 10^8 PFU/mL were administered every 3 weeks for up to 35 cycles in total. Participants also received pembrolizumab at a dose of 200 mg as an IV infusion every 3 weeks for up to 35 cycles.
- Cohort 4 - Adjuvant Setting - Disease Free Interval ≥ 6 Months: Included participants who received anti PD-1 therapy in the adjuvant setting and experienced confirmed disease progression following a disease-free interval of ≥ 6 months after starting the adjuvant PD-1 inhibitor.
  Participants received talimogene laherparepvec at an initial dose of up to 4.0 mL of 10^6 PFU/mL by intralesional injection into injectable cutaneous, subcutaneous and nodal legions on Day 1. Subsequent doses of up to 4.0 mL of 10^8 PFU/mL were administered every 3 weeks for up to 35 cycles in total. Participants also received pembrolizumab at a dose of 200 mg as an IV infusion every 3 weeks for up to 35 cycles.
Period: Overall Study
Arm/Group | Cohort 1 - Locally Recurrent/Metastatic - Primary Resistance | Cohort 2 - Locally Recurrent/Metastatic - Acquired Resistance | Cohort 3 - Adjuvant Setting - Disease Free Interval < 6 Months | Cohort 4 - Adjuvant Setting - Disease Free Interval ≥ 6 Months
Started | 27 | 15 | 15 | 15
Received Talimogene Laherparepvec | 26 | 15 | 15 | 15
Received Pembrolizumab | 26 | 15 | 15 | 15
Completed | 6 | 3 | 11 | 8
Not Completed | 21 | 12 | 4 | 7
Not completed — Death | 17 | 12 | 4 | 7
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Withdrawal of consent from study | 3 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: All enrolled participants who received at least 1 dose of talimogene laherparepvec or pembrolizumab.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 - Locally Recurrent/Metastatic - Primary Resistance | Cohort 2 - Locally Recurrent/Metastatic - Acquired Resistance | Cohort 3 - Adjuvant Setting - Disease Free Interval < 6 Months | Cohort 4 - Adjuvant Setting - Disease Free Interval ≥ 6 Months | Total
Number analyzed (Participants) | 26 | 15 | 15 | 15 | 71
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.2 (14.6) | 65.5 (13.2) | 59.4 (13.0) | 63.5 (10.3) | 62.9 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 5 | 2 | 23
  Male | 18 | 7 | 10 | 13 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 25 | 14 | 14 | 15 | 68
  Unknown or Not Reported | 1 | 1 | 1 | 0 | 3
Race [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Black (or African American) | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  White | 25 | 14 | 14 | 15 | 68
  Other | 1 | 1 | 1 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) Per Modified RECIST v1.1
Description: ORR was defined as the incidence of a best overall response (BOR) of complete response (CR) or partial response (PR) per modified RECIST v1.1:
  * CR: Disappearance of all target and non-target lesions. Any pathological lymph nodes (whether target or non-target) must have had a reduction in short axis to < 10 mm. All lymph nodes must have been non-pathological in size (< 10mm short axis).
  * PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  * Non-CR/Non-progressive disease (PD): Persistence of 1 or more non-target lesion(s).
Time Frame: Every 12 weeks. Maximum overall time on-study (treatment + follow up) was 46.23 months
Population: Full Analysis Set: Includes all enrolled participants who have received at least 1 dose of talimogene laherparepvec and 1 dose of pembrolizumab in combination.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort 1 - Locally Recurrent/Metastatic - Primary Resistance | Cohort 2 - Locally Recurrent/Metastatic - Acquired Resistance | Cohort 3 - Adjuvant Setting - Disease Free Interval < 6 Months | Cohort 4 - Adjuvant Setting - Disease Free Interval ≥ 6 Months
Number analyzed (Participants) | 26 | 15 | 15 | 15
Percentage of Participants | 3.8 [0.10 to 19.64] | 6.7 [0.17 to 31.95] | 40.0 [16.34 to 67.71] | 46.7 [21.27 to 73.41]

2. Secondary Outcome: Complete Response Rate (CRR) Per Modified RECIST v1.1
Description: CRR was defined as the incidence of a BOR of CR per modified RECIST v1.1:
  * CR: Disappearance of all target and non-target lesions. Any pathological lymph nodes (whether target or non-target) must have had a reduction in short axis to < 10 mm. All lymph nodes must have been non-pathological in size (< 10mm short axis).
  Confirmation of CR was not required per modified RECIST v1.1.
Time Frame: Every 12 weeks. Maximum overall time on-study (treatment + follow up) was 46.23 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort 1 - Locally Recurrent/Metastatic - Primary Resistance | Cohort 2 - Locally Recurrent/Metastatic - Acquired Resistance | Cohort 3 - Adjuvant Setting - Disease Free Interval < 6 Months | Cohort 4 - Adjuvant Setting - Disease Free Interval ≥ 6 Months
Number analyzed (Participants) | 26 | 15 | 15 | 15
Percentage of Participants | 0 [NA to NA] — No participants achieved a CR so the 95% confidence interval was not estimable. | 0 [NA to NA] — No participants achieved a CR so the 95% confidence interval was not estimable. | 20.0 [4.33 to 48.09] | 20.0 [4.33 to 48.09]

3. Secondary Outcome: Complete Response Rate (iCRR) Per Modified Immune-related Response Criteria (irRC) RECIST v1.1
Description: iCRR was defined as the incidence of a best overall response (iBOR) of a complete response (iCR) per modified irRC-RECIST:
  * iCR: Disappearance of all lesions (whether measurable or not and whether baseline or new). Any pathological lymph nodes (whether target or nontarget) must have had a reduction in short axis to < 10 mm.
  Confirmation of iCR was required per modified irRC-RECIST.
Time Frame: Every 12 weeks. Maximum overall time on-study (treatment + follow up) was 46.23 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort 1 - Locally Recurrent/Metastatic - Primary Resistance | Cohort 2 - Locally Recurrent/Metastatic - Acquired Resistance | Cohort 3 - Adjuvant Setting - Disease Free Interval < 6 Months | Cohort 4 - Adjuvant Setting - Disease Free Interval ≥ 6 Months
Number analyzed (Participants) | 26 | 15 | 15 | 15
Percentage of Participants | 0 [NA to NA] — No participants achieved an iCR so the 95% confidence interval is not evaluable. | 0 [NA to NA] — No participants achieved an iCR so the 95% confidence interval is not evaluable. | 26.7 [7.79 to 55.10] | 20.0 [4.33 to 48.09]

4. Secondary Outcome: BOR Per Modified RECIST v1.1
Description: BOR was the best overall visit response up to & including the first overall visit response of PD:
  * CR: Disappearance of all target & non-target lesions. Any pathological lymph nodes must have had a reduction in short axis to <10 mm. All lymph nodes must have been non-pathological in size.
  * PR: ≥30% decrease in the sum of diameters of target lesions.
  * Stable disease (SD): Neither sufficient shrinkage to qualify for PR/CR nor sufficient increase to qualify for PD.
  * PD: ≥20% increase in the sum of diameters of target lesions and an increase of ≥5mm. Progression of existing non-target lesions.
  * Unable to evaluate (UE): Any lesion present at baseline which was not assessed or unable to be evaluated leading to an inability to determine the status of that particular tumor.
  * Non-CR/Non-PD: Persistence of 1+ non-target lesion(s). Non-CR/non-PD was relevant to participants who did not have measurable disease at baseline.
  Confirmation of CR, PR & PD were not required per modified RECIST 1.1.
Time Frame: Every 12 weeks. Maximum overall time on-study (treatment + follow up) was 46.23 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - Locally Recurrent/Metastatic - Primary Resistance | Cohort 2 - Locally Recurrent/Metastatic - Acquired Resistance | Cohort 3 - Adjuvant Setting - Disease Free Interval < 6 Months | Cohort 4 - Adjuvant Setting - Disease Free Interval ≥ 6 Months
Number analyzed (Participants) | 26 | 15 | 15 | 15
Participants
  CR | 0 | 0 | 3 | 3
  PR | 1 | 1 | 3 | 4
  SD | 7 | 4 | 0 | 6
  PD | 11 | 5 | 9 | 1
  UE | 0 | 1 | 0 | 0
  Non-CR/Non-PD | 1 | 0 | 0 | 0
  Not Done | 6 | 4 | 0 | 1

5. Secondary Outcome: Best Overall Response (iBOR) Per Modified irRC-RECIST
Description: iBOR was defined as the best overall visit response up to and including the first overall visit response of progressive disease (iPD) per modified irRC-RECIST:
  * iCR: Disappearance of all lesions (whether measurable or not and whether baseline or new). Any pathological lymph nodes (whether target or nontarget) must have a reduction in short axis to < 10 mm.
  * Partial response (iPR): Decrease in tumor burden ≥ 30% relative to baseline.
  * Stable disease (iSD): Neither sufficient shrinkage to qualify for iPR or iCR nor sufficient increase to qualify for iPD.
  * iPD: Increase in tumor burden ≥ 20% and at least 5 mm absolute increase.
  * Unable to evaluate (iUE): Any lesion present at baseline or a new measurable lesion which was not assessed or was unable to be evaluated leading to an inability to determine the status of that particular tumor for that time point.
  Confirmation of iCR, iPR and iPD was required per modified irRC-RECIST.
Time Frame: Every 12 weeks. Maximum overall time on-study (treatment + follow up) was 46.23 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - Locally Recurrent/Metastatic - Primary Resistance | Cohort 2 - Locally Recurrent/Metastatic - Acquired Resistance | Cohort 3 - Adjuvant Setting - Disease Free Interval < 6 Months | Cohort 4 - Adjuvant Setting - Disease Free Interval ≥ 6 Months
Number analyzed (Participants) | 26 | 15 | 15 | 15
Participants
  iCR | 0 | 0 | 4 | 3
  iPR | 3 | 1 | 7 | 4
  iSD | 10 | 5 | 0 | 6
  iPD | 5 | 4 | 1 | 0
  iUE | 2 | 1 | 2 | 1
  Not Done | 6 | 4 | 1 | 1

6. Secondary Outcome: Durable Response Rate (DRR) Per Modified RECIST v1.1
Description: DRR was defined as the percentage of participants with a CR or PR per modified RECIST v1.1 with a duration of response (DOR) ≥ 6 months. One month was calculated based on 365.25 days per year.
  * CR: Disappearance of all target and non-target lesions. Any pathological lymph nodes (whether target or non-target) must have had a reduction in short axis to < 10 mm. All lymph nodes must have been non-pathological in size (< 10mm short axis).
  * PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  Confirmation of CR and PR were not required per modified RECIST v1.1.
Time Frame: Every 12 weeks. Maximum overall time on-study (treatment + follow up) was 46.23 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort 1 - Locally Recurrent/Metastatic - Primary Resistance | Cohort 2 - Locally Recurrent/Metastatic - Acquired Resistance | Cohort 3 - Adjuvant Setting - Disease Free Interval < 6 Months | Cohort 4 - Adjuvant Setting - Disease Free Interval ≥ 6 Months
Number analyzed (Participants) | 26 | 15 | 15 | 15
Percentage of Participants | 3.8 [0.10 to 19.64] | 6.7 [0.17 to 31.95] | 40.0 [16.34 to 67.71] | 26.7 [7.79 to 55.10]

7. Secondary Outcome: Durable Response Rate (iDRR) Per Modified irRC-RECIST
Description: iDRR was defined as the percentage of participants with an iCR or iPR per modified irRC-RECIST with a duration of response (iDOR) ≥ 6 months. One month was calculated based on 365.25 days per year.
  * iCR: Disappearance of all lesions (whether measurable or not and whether baseline or new). Any pathological lymph nodes (whether target or nontarget) must have a reduction in short axis to < 10 mm.
  * iPR: Decrease in tumor burden ≥ 30% relative to baseline.
  Confirmation of iCR and iPR were required per modified irRC-RECIST.
Time Frame: Every 12 weeks. Maximum overall time on-study (treatment + follow up) was 46.23 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort 1 - Locally Recurrent/Metastatic - Primary Resistance | Cohort 2 - Locally Recurrent/Metastatic - Acquired Resistance | Cohort 3 - Adjuvant Setting - Disease Free Interval < 6 Months | Cohort 4 - Adjuvant Setting - Disease Free Interval ≥ 6 Months
Number analyzed (Participants) | 26 | 15 | 15 | 15
Percentage of Participants | 11.5 [2.45 to 30.15] | 6.7 [0.17 to 31.95] | 73.3 [44.90 to 92.21] | 40.0 [16.34 to 67.71]

8. Secondary Outcome: DOR Per Modified RECIST v1.1
Description: DOR was defined as the time from the date of an initial response of CR or PR to the earlier of PD/death. Participants who had not ended their response at the time of analysis were censored at their last evaluable tumor assessment date before start of first subsequent anticancer therapy. One month was calculated based on 365.25 days per year.
  * CR:Disappearance of all target & non-target lesions. All lymph nodes must have a reduction in short axis to <10 mm. Any pathological lymph nodes must have had a reduction in short axis to <10 mm. All lymph nodes must have been non-pathological in size (<10mm short axis).
  * PR:At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  * PD:At least a 20% increase in the sum of diameters of target lesions. The sum must also demonstrate an increase of at least 5mm. Unequivocal progression of existing non-target lesions.
  Confirmation of CR, PR and PD were not required per modified RECIST v1.1.
Time Frame: Every 12 weeks. Maximum overall time on-study (treatment + follow up) was 46.23 months
Population: Full Analysis Set: Includes all enrolled participants who have received at least 1 dose of talimogene laherparepvec and 1 dose of pembrolizumab in combination. Only participants who had an initial response of CR or PR were included.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1 - Locally Recurrent/Metastatic - Primary Resistance | Cohort 2 - Locally Recurrent/Metastatic - Acquired Resistance | Cohort 3 - Adjuvant Setting - Disease Free Interval < 6 Months | Cohort 4 - Adjuvant Setting - Disease Free Interval ≥ 6 Months
Number analyzed (Participants) | 1 | 1 | 6 | 7
Months | 22.768 [NA to NA] — Dispersion data could not be calculated as only 1 participant experienced a response. | 7.655 [NA to NA] — Dispersion data could not be calculated as only 1 participant experienced a response. | NA [19.351 to NA] — Median DOR and upper limit of 95% confidence interval was not reached due to the low number of events (PD or death). | 13.700 [5.520 to NA] — Upper limit of 95% confidence interval was not reached due to the low number of events (PD or death).

9. Secondary Outcome: iDOR Per Modified irRC-RECIST
Description: iDOR was defined as the time from the date of an initial response that is subsequently confirmed to the earlier of iPD per modified irRC-RECIST.
  Participants who had not ended their response at the time of analysis were censored at their last evaluable tumor assessment date before start of first subsequent anticancer therapy. One month was calculated based on 365.25 days per year.
  * iCR: Disappearance of all target and non-target lesions. All lymph nodes must have a reduction in short axis to < 10 mm.
  * iPR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  * iPD: At least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5mm. Unequivocal progression of existing non-target lesions.
Time Frame: Every 12 weeks. Maximum overall time on-study (treatment + follow up) was 46.23 months
Population: Full Analysis Set: Includes all enrolled participants who have received at least 1 dose of talimogene laherparepvec and 1 dose of pembrolizumab in combination. Only participants who had an initial response of iCR or iPR were included.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1 - Locally Recurrent/Metastatic - Primary Resistance | Cohort 2 - Locally Recurrent/Metastatic - Acquired Resistance | Cohort 3 - Adjuvant Setting - Disease Free Interval < 6 Months | Cohort 4 - Adjuvant Setting - Disease Free Interval ≥ 6 Months
Number analyzed (Participants) | 3 | 1 | 11 | 7
Months | NA [22.768 to NA] — Median iDOR and upper limit of 95% confidence interval was not reached due to the low number of events (PD or death). | 7.655 [NA to NA] — Dispersion data could not be calculated as only 1 participant experienced a response. | NA [NA to NA] — No participants experienced a response that had ended so no data were estimable | NA [11.302 to NA] — Median iDOR and upper limit of 95% confidence interval was not reached due to the low number of events (PD or death).

10. Secondary Outcome: Disease Control Rate (DCR) Per Modified RECIST v1.1
Description: DCR per modified RECIST v1.1 was defined as the incidence of a BOR of CR, PR or SD.
  * CR: Disappearance of all target and non-target lesions. Any pathological lymph nodes (whether target or non-target) must have had a reduction in short axis to < 10 mm. All lymph nodes must have been non-pathological in size (< 10mm short axis
  * PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  * SD: Neither sufficient shrinkage to qualify for PR or CR nor sufficient increase to qualify for PD.
  Confirmation of CR and PR were not required per modified RECIST v1.1.
Time Frame: Every 12 weeks. Maximum overall time on-study (treatment + follow up) was 46.23 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort 1 - Locally Recurrent/Metastatic - Primary Resistance | Cohort 2 - Locally Recurrent/Metastatic - Acquired Resistance | Cohort 3 - Adjuvant Setting - Disease Free Interval < 6 Months | Cohort 4 - Adjuvant Setting - Disease Free Interval ≥ 6 Months
Number analyzed (Participants) | 26 | 15 | 15 | 15
Percentage of Participants | 30.8 [14.33 to 51.79] | 33.3 [11.82 to 61.62] | 40.0 [16.34 to 67.71] | 86.7 [59.54 to 98.34]

11. Secondary Outcome: Disease Control Rate (iDCR) Per Modified irRC-RECIST
Description: iDCR per modified irRC-RECIST was defined as the incidence of an iBOR of iCR, iPR or iSD.
  * iCR: Disappearance of all target and non-target lesions. All lymph nodes must have a reduction in short axis to < 10 mm.
  * iPR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  * iSD: Neither sufficient shrinkage to qualify for iPR or iCR nor sufficient increase to qualify for iPD.
  Confirmation of iCR and iPR were required per modified irRC-RECIST.
Time Frame: Every 12 weeks. Maximum overall time on-study (treatment + follow up) was 46.23 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort 1 - Locally Recurrent/Metastatic - Primary Resistance | Cohort 2 - Locally Recurrent/Metastatic - Acquired Resistance | Cohort 3 - Adjuvant Setting - Disease Free Interval < 6 Months | Cohort 4 - Adjuvant Setting - Disease Free Interval ≥ 6 Months
Number analyzed (Participants) | 26 | 15 | 15 | 15
Percentage of Participants | 50.0 [29.93 to 70.07] | 40.0 [16.34 to 67.71] | 73.3 [44.90 to 92.21] | 86.7 [59.54 to 98.34]

12. Secondary Outcome: Objective Response Rate (iORR) Per Modified irRC-RECIST
Description: iORR was defined as the incidence of an iBOR of iCR or iPR per modified irRC-RECIST
  * iCR: Disappearance of all lesions (whether measurable or not and whether baseline or new). Any pathological lymph nodes (whether target or nontarget) must have a reduction in short axis to < 10 mm.
  * iPR: Decrease in tumor burden ≥ 30% relative to baseline.
  Confirmation of iCR and iPR were required per modified irRC-RECIST.
Time Frame: Every 12 weeks. Maximum overall time on-study (treatment + follow up) was 46.23 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort 1 - Locally Recurrent/Metastatic - Primary Resistance | Cohort 2 - Locally Recurrent/Metastatic - Acquired Resistance | Cohort 3 - Adjuvant Setting - Disease Free Interval < 6 Months | Cohort 4 - Adjuvant Setting - Disease Free Interval ≥ 6 Months
Number analyzed (Participants) | 26 | 15 | 15 | 15
Percentage of Participants | 11.5 [2.45 to 30.15] | 6.7 [0.17 to 31.95] | 73.3 [44.90 to 92.21] | 46.7 [21.27 to 73.41]

13. Secondary Outcome: Progression Free Survival (PFS) Per Modified RECIST v1.1
Description: PFS per modified RECIST 1.1 was defined as the interval from first dose to the earlier event of PD or death from any cause. Participants without an event were censored at their last evaluable post-baseline tumor assessment if available, otherwise were censored on study Day 1. One month was calculated based on 365.25 days per year.
  - PD: At least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5mm. Unequivocal progression of existing non-target lesions.
Time Frame: Every 12 weeks. Maximum overall time on-study (treatment + follow up) was 46.23 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1 - Locally Recurrent/Metastatic - Primary Resistance | Cohort 2 - Locally Recurrent/Metastatic - Acquired Resistance | Cohort 3 - Adjuvant Setting - Disease Free Interval < 6 Months | Cohort 4 - Adjuvant Setting - Disease Free Interval ≥ 6 Months
Number analyzed (Participants) | 26 | 15 | 15 | 15
Months | 3.614 [2.793 to 5.520] | 4.830 [2.431 to 13.207] | 2.793 [2.661 to 27.433] | 13.897 [5.552 to 19.318]

14. Secondary Outcome: Progression Free Survival (iPFS) Per Modified irRC-RECIST
Description: iPFS per modified irRC-RECIST was defined as the interval from first dose to the earlier event of iPD or death from any cause. Participants without an event were censored at their last evaluable post-baseline tumor assessment if available, otherwise were censored on study Day 1. One month was calculated based on 365.25 days per year.
  - iPD: Increase in tumor burden ≥ 20% and at least 5 mm absolute increase.
Time Frame: Every 12 weeks. Maximum overall time on-study (treatment + follow up) was 46.23 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1 - Locally Recurrent/Metastatic - Primary Resistance | Cohort 2 - Locally Recurrent/Metastatic - Acquired Resistance | Cohort 3 - Adjuvant Setting - Disease Free Interval < 6 Months | Cohort 4 - Adjuvant Setting - Disease Free Interval ≥ 6 Months
Number analyzed (Participants) | 26 | 15 | 15 | 15
Months | 6.899 [2.793 to 25.232] | 8.214 [2.694 to 15.014] | NA [2.694 to NA] — Median and upper limit of the 95% confidence limit were not estimable due to the low number of events (iPD or death). | 25.955 [16.756 to NA] — Upper limit of the 95% confidence limit was not estimable due to the low number of events (iPD or death).

15. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the interval from first dose to death from any cause. Participants without an event were censored at the last date known to be alive. One month was calculated based on 365.25 days per year.
Time Frame: Every 12 weeks. Maximum overall time on-study (treatment + follow up) was 46.23 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1 - Locally Recurrent/Metastatic - Primary Resistance | Cohort 2 - Locally Recurrent/Metastatic - Acquired Resistance | Cohort 3 - Adjuvant Setting - Disease Free Interval < 6 Months | Cohort 4 - Adjuvant Setting - Disease Free Interval ≥ 6 Months
Number analyzed (Participants) | 26 | 15 | 15 | 15
Months | 24.608 [6.538 to 42.086] | 15.014 [2.760 to 38.374] | NA [8.575 to NA] — Median and upper limit of the 95% confidence interval were not estimable due to the low number of events. | NA [20.370 to NA] — Median and upper limit of the 95% confidence interval were not estimable due to the low number of events.

16. Secondary Outcome: Number of Participants Who Experienced a Treatment-emergent Adverse Event (TEAE)
Description: Evaluation of TEAEs included the number of participants with at least 1:
  * TEAE
  * Treatment-related TEAE
  * Common Terminology Criteria for Adverse Events (CTCAE) grade ≥ 3 TEAE
  * Treatment-related CTCAE grade ≥ 3 TEAE
  * Serious TEAE
  * Serious treatment-related TEAE
  * Fatal TEAE
  * Fatal treatment-related TEAE
  * TEAE of interest
  Serious TEAEs were collected up to 90 days post-last dose of treatment. Non-serious TEAEs were collected up to 30 days post-last dose of treatment.
  A CTCAE grade ≥ 3 was determined using the CTCAE grading systems based on CTCAE version 5.0 per the below definitions:
  * Grade 3: Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care activities of daily living.
  * Grade 4: Life-threatening consequences; urgent intervention indicated.
  * Grade 5: Death related to TEAE.
  Abnormal laboratory tests were also recorded as TEAEs.
Time Frame: Serious TEAEs were collected up to 90 days post-last dose of treatment. Non-serious TEAEs were collected up to 30 days post-last dose of treatment. The maximum duration of treatment exposure was 105.9 weeks.
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - Locally Recurrent/Metastatic - Primary Resistance | Cohort 2 - Locally Recurrent/Metastatic - Acquired Resistance | Cohort 3 - Adjuvant Setting - Disease Free Interval < 6 Months | Cohort 4 - Adjuvant Setting - Disease Free Interval ≥ 6 Months
Number analyzed (Participants) | 26 | 15 | 15 | 15
Participants
  TEAEs | 24 | 15 | 15 | 14
  Treatment-related TEAEs | 17 | 10 | 14 | 13
  CTCAE Grade ≥ 3 TEAEs | 11 | 8 | 4 | 8
  CTCAE Grade ≥ 3 Treatment-related TEAEs | 2 | 3 | 0 | 6
  Serious TEAEs | 12 | 7 | 4 | 7
  Serious Treatment-related TEAEs | 1 | 2 | 0 | 3
  Fatal TEAEs | 5 | 3 | 1 | 3
  Fatal Treatment-related TEAEs | 0 | 0 | 0 | 1
  TEAEs of Interest | 21 | 14 | 15 | 14

17. Secondary Outcome: Time to First Subsequent Anti-cancer Therapy
Description: Time to first subsequent anti-cancer therapy was defined as the time from enrollment to the start of subsequent anticancer therapy. Participants who did not start subsequent anticancer therapy were censored as the last known to be alive date. One month was calculated based on 365.25 days per year.
Time Frame: Every 12 weeks. Maximum overall time on-study (treatment + follow up) was 46.23 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1 - Locally Recurrent/Metastatic - Primary Resistance | Cohort 2 - Locally Recurrent/Metastatic - Acquired Resistance | Cohort 3 - Adjuvant Setting - Disease Free Interval < 6 Months | Cohort 4 - Adjuvant Setting - Disease Free Interval ≥ 6 Months
Number analyzed (Participants) | 26 | 15 | 15 | 15
Months | 11.466 [6.209 to 38.111] | 7.852 [2.793 to NA] — Upper limit of the 95% confidence interval was not estimable due to the low number of participants who received subsequent anti-cancer therapy. | NA [25.758 to NA] — Median and upper limit of the 95% confidence interval were not estimable due to the low number of participants who received subsequent anti-cancer therapy. | 23.097 [11.532 to NA] — Upper limit of the 95% confidence interval was not estimable due to the low number of participants who received subsequent anti-cancer therapy.

ADVERSE EVENTS:
Time Frame: Serious TEAEs were collected up to 90 days post-last dose of treatment. Non-serious TEAEs were collected up to 30 days post-last dose of treatment. The maximum duration of treatment exposure was 105.9 weeks.
Description: All-cause mortality was collected for all enrolled participants. Serious TEAEs and non-serious TEAEs were collected for the safety analysis set which included all enrolled participants who received at least 1 dose of talimogene laherparepvec or pembrolizumab.
Groups:
- Cohort 1 - Locally Recurrent/Metastatic - Primary Resistance: Included participants who received anti-PD-1 therapy in the locally recurrent/metastatic setting and experienced a best overall response of disease progression or stable disease prior to confirmed disease progression. Participants received talimogene laherparepvec at an initial dose of up to 4.0 mL of 10^6 PFU/mL by intralesional injection into injectable cutaneous, subcutaneous and nodal legions on Day 1. Subsequent doses of up to 4.0 mL of 10^8 PFU/mL were administered every 3 weeks for up to 35 cycles in total. Participants also received pembrolizumab at a dose of 200 mg as an IV infusion every 3 weeks for up to 35 cycles.
Arm/Group | Cohort 1 - Locally Recurrent/Metastatic - Primary Resistance | Cohort 2 - Locally Recurrent/Metastatic - Acquired Resistance | Cohort 3 - Adjuvant Setting - Disease Free Interval < 6 Months | Cohort 4 - Adjuvant Setting - Disease Free Interval ≥ 6 Months
All-Cause Mortality (participants affected / at risk) | 17/27 | 12/15 | 4/15 | 7/15
Serious Adverse Events (participants affected / at risk) | 12/26 | 7/15 | 4/15 | 7/15
Other Adverse Events (participants affected / at risk) | 20/26 | 15/15 | 15/15 | 14/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 - Locally Recurrent/Metastatic - Primary Resistance (N=26) | Cohort 2 - Locally Recurrent/Metastatic - Acquired Resistance (N=15) | Cohort 3 - Adjuvant Setting - Disease Free Interval < 6 Months (N=15) | Cohort 4 - Adjuvant Setting - Disease Free Interval ≥ 6 Months (N=15)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0 | 0
Adrenocortical insufficiency acute (Endocrine disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Intussusception (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Death (General disorders) | 0 | 0 | 0 | 2
General physical health deterioration (General disorders) | 2 | 1 | 0 | 0
Liver injury (Hepatobiliary disorders) | 1 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 1 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 1 | 1
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Brain oedema (Nervous system disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0
Renal disorder (Renal and urinary disorders) | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hypophysitis (Endocrine disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 - Locally Recurrent/Metastatic - Primary Resistance (N=26) | Cohort 2 - Locally Recurrent/Metastatic - Acquired Resistance (N=15) | Cohort 3 - Adjuvant Setting - Disease Free Interval < 6 Months (N=15) | Cohort 4 - Adjuvant Setting - Disease Free Interval ≥ 6 Months (N=15)
Anaemia (Blood and lymphatic system disorders) | 4 | 2 | 1 | 2
Anaemia vitamin B12 deficiency (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Eosinophilia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0 | 1
Conjunctival suffusion (Eye disorders) | 0 | 1 | 0 | 0
Diplopia (Eye disorders) | 0 | 1 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 1
Retinal disorder (Eye disorders) | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0
Xerophthalmia (Eye disorders) | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 2 | 0
Anal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0 | 2 | 2
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 2 | 2 | 7
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 6 | 4 | 3 | 3
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 4 | 2 | 0 | 2
Asthenia (General disorders) | 3 | 1 | 2 | 2
Axillary pain (General disorders) | 0 | 1 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 1
Chills (General disorders) | 6 | 2 | 2 | 2
Face oedema (General disorders) | 0 | 0 | 1 | 0
Fatigue (General disorders) | 4 | 5 | 6 | 5
Hyperthermia (General disorders) | 0 | 1 | 2 | 0
Influenza like illness (General disorders) | 2 | 1 | 7 | 2
Injection site extravasation (General disorders) | 0 | 0 | 1 | 0
Injection site haemorrhage (General disorders) | 0 | 0 | 1 | 1
Injection site inflammation (General disorders) | 0 | 1 | 0 | 0
Injection site oedema (General disorders) | 0 | 0 | 1 | 0
Injection site pain (General disorders) | 3 | 2 | 4 | 1
Injection site paraesthesia (General disorders) | 0 | 1 | 0 | 0
Injection site reaction (General disorders) | 0 | 0 | 2 | 0
Pain (General disorders) | 2 | 0 | 0 | 3
Peripheral swelling (General disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 7 | 6 | 5 | 7
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hepatic cytolysis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Contrast media allergy (Immune system disorders) | 0 | 0 | 0 | 1
Sarcoidosis (Immune system disorders) | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0
Cellulitis orbital (Infections and infestations) | 0 | 0 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 1
Diarrhoea infectious (Infections and infestations) | 0 | 0 | 0 | 1
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 0 | 1
Genital herpes simplex (Infections and infestations) | 0 | 0 | 1 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 1 | 0
Herpes simplex reactivation (Infections and infestations) | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 2 | 1
Skin infection (Infections and infestations) | 0 | 0 | 1 | 0
Tinea versicolour (Infections and infestations) | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Wound infection (Infections and infestations) | 0 | 1 | 0 | 0
Accident at home (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1 | 2
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 1 | 1
Blood creatinine increased (Investigations) | 2 | 1 | 0 | 1
Blood pressure increased (Investigations) | 0 | 1 | 0 | 0
Blood thyroid stimulating hormone increased (Investigations) | 1 | 1 | 1 | 0
Body temperature increased (Investigations) | 0 | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 0
Lipase increased (Investigations) | 0 | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 1
Transaminases increased (Investigations) | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 2 | 1 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 3 | 0 | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 2 | 4
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 4 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 4 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 3 | 2 | 2
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Rheumatic disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 2 | 5 | 1
Lethargy (Nervous system disorders) | 0 | 0 | 2 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 2 | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 1 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 0 | 0 | 1
Sleep disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urethral dilatation (Renal and urinary disorders) | 0 | 1 | 0 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hair colour changes (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 5 | 2
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 4 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Scab (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin hyperplasia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Umbilical discharge (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Vitiligo (Skin and subcutaneous tissue disorders) | 2 | 3 | 1 | 2
Skin neoplasm excision (Surgical and medical procedures) | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 1 | 0 | 0 | 2
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0 | 1 | 0
Hypophysitis (Endocrine disorders) | 0 | 0 | 0 | 1
Change of bowel habit (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 1 | 0 | 1 | 0
Xerosis (General disorders) | 0 | 0 | 1 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 1 | 0
COVID-19 (Infections and infestations) | 1 | 1 | 2 | 0
Cystitis (Infections and infestations) | 2 | 0 | 0 | 0
Dermatophytosis (Infections and infestations) | 0 | 0 | 1 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 1
Mastoiditis (Infections and infestations) | 0 | 1 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 1 | 0 | 0
Vaginal infection (Infections and infestations) | 0 | 0 | 1 | 0
Immunisation reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Skin wound (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Tumour fistulisation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0
Penile dermatitis (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Lichen planus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2021-06-09): https://cdn.clinicaltrials.gov/large-docs/81/NCT04068181/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-12): https://cdn.clinicaltrials.gov/large-docs/81/NCT04068181/SAP_001.pdf